CLINICAL TRIAL: NCT05967572
Title: The Effect of Different Music Listened During Retinopathy Examination to Premature Infants on Their Pain and Comfort Level: A Randomized Controlled Trial
Brief Title: The Effect of Different Music Listened During Retinopathy Examination to Premature Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Semra Kose, Asisstant Proffessor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NecmettinEUSKose
Record Dates: First submitted 2023-07-08; First posted 2023-08-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Retinopathy of Prematurity; Newborn
Keywords: Pain; Nursing; Comfort; Music; Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity; Pain; Premature Birth

STUDY DESIGN:
Intervention Model Description: The research is a stratified randomized controlled experimental type study.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Behavioral responses and physiological measurements of premature babies will be evaluated by using these video recordings by the nurse responsible for ROP, a lecturer who specializes in newborns and pain, and the researcher (3 experts), who are experienced in the ROP examination who do not know the groups, and who waive all rights of the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experiment 1 (Rainstick) (Experimental): The experimental group will start playing music 3 minutes before the start of the process. The examination begins with the insertion of the speculum into the eye. The duration of the examination depends on the visibility of the vascularity in the retina and the examination will end with the removal of the speculum from the eye. The rain bar will continue to play during the ROP inspection. The rain stick will be played 25cm away from the baby.
  Interventions: Other: Research processes;
- Experiment 2 (Music-The Happiest Baby) (Experimental): During the ROP examination, Dr. Harvery Karp's "The Happiest Baby", which consists of only intrauterine sounds, is a group of babies who are listened to. The experimental group will start playing music 3 minutes before the start of the process. The examination begins with the insertion of the speculum into the eye. The duration of the examination depends on the visibility of the vascularity in the retina and the examination will end with the removal of the speculum from the eye. Music will continue to play during the ROP exam. The voice recorder that will play The Happiest Baby will be placed 25 cm away from the baby. In the study, the music volume will be set as 45-50 decibels.
  Interventions: Other: Research processes;
- Control (No Intervention): It is the group of infants who receive routine care during the ROP examination. In the control group, a routine ROP procedure will be performed without any music before, during and after the ROP examination.

INTERVENTIONS:
Other: Research processes; — 1. Before Inspection: information will be obtained and premature babies will be monitored by wearing a pulse oximeter device and their heart rate and oxygen saturation value will be recorded for control purposes. By making video recordings of each premature baby; PIPP pain score, PBIC comfort score, control oxygen saturation and peak heart rate values will be recorded 3 minutes before the ROP examination. Babies will be fed and changed at least half an hour before the examination.
  2. Inspection Sequence: PIPP pain score, PBIC comfort score, control oxygen saturation and peak heart rate values will be recorded and evaluated from the video recording that continues with the start of the examination.
  3. End of Inspection: Infants whose both eye examinations are completed and whose monitoring and video recording continue will be recorded and evaluated 3 minutes after the end of the examination, with PIPP pain score, PBIC comfort score, control oxygen saturation and heart rate values.
  Arms: Experiment 1 (Rainstick); Experiment 2 (Music-The Happiest Baby)

SUMMARY:
Retinopathy of Prematurity (ROP); It is a disease of premature and low birth weight infants, characterized by incomplete vascularization of the retina, etiology and pathogenesis of which is unknown, and causes vision loss. There is an increase in the incidence and severity of ROP development in direct proportion to the decrease in birth week and birth weight. While ROP is a problem below 32 weeks of gestation in developed countries, it is reported to develop severely up to 34 weeks of gestation in developing countries. In a multicenter study conducted by the Turkish Neonatology Society in our country, the frequency of ROP in very low birth weight preterm infants was found to be 42%, and the frequency of advanced ROP was 11%. The incidence of ROP in babies with a gestational age of 33-35 weeks was 6.1%, and advanced ROP was 6 per thousand. The frequency of ROP was found to be 10.3% in babies with a birth weight of 1500-2000 grams, and severe ROP was reported in 19 of these babies. ROP examination is a procedure that causes pain, deterioration in comfort and physiological changes in preterm newborns. After this examination, an increase in blood pressure and heart rate and a decrease in oxygen saturation are observed. Pharmacological and non-pharmacological (non-pharmacological) methods are used to reduce the pain and increase the comfort level of the premature newborn. As a pharmacological method, there is no other routine method used to reduce pain other than the administration of local anesthetic drops before the examination. Because of this situation, nurses apply various non-pharmacological methods to alleviate pain. These methods are; breast milk, sucrose use, oral dextrose use, non-nutritive sucking, positioning, listening to music and mother's voice. In the literature, no specific study was found in which music was used to reduce pain and increase the comfort level during the ROP examination. Therefore, this research will be carried out to determine the effect of different music played on the pain and comfort level of premature babies during the retinopathy examination.

DETAILED DESCRIPTION:
Retinopathy of Prematurity (ROP); It is a disease characterized by incomplete vascularization of the retina seen in premature and low birth weight infants, the etiology and pathogenesis of which are unknown, causing vision loss. There is an increase in the incidence and severity of ROP development in direct proportion to the decrease in the week of birth and birth weight. While ROP is a problem below 32 weeks of gestation in developed countries, it is reported to develop severely up to 34 weeks of gestation in developing countries. In a multicenter study conducted by the Turkish Neonatology Society in our country, the frequency of ROP in very low birth weight preterm infants was found to be 42%, and the frequency of advanced ROP was 11%. The incidence of ROP in babies with a gestational age of 33-35 weeks was 6.1%, and advanced ROP was 6 per thousand. The frequency of ROP was found to be 10.3% in babies with a birth weight of 1500-2000 grams, and severe ROP was reported in 19 of these babies. Thanks to the increasing frequency of preterm birth in recent years and scientific and technological advances in neonatology, life expectancy is extended up to the 23rd week of gestation. However, this increased the incidence of retinopathy. Therefore, it is of great importance for neotologists, pediatricians and nurses who care for preterms to know the pathophysiology, staging, risk factors and principles of appropriate care for them in reducing the incidence, possible complications and mortality rates of ROP. ROP examination is a procedure that causes pain, deterioration in comfort and physiological changes in preterm newborns. After this examination, an increase in blood pressure and heart rate and a decrease in oxygen saturation are observed. These physiological changes observed after the examination continue for 24 hours. Pharmacological and non-pharmacological (non-pharmacological) methods are used to reduce the pain and increase the comfort level of the premature newborn. As a pharmacological method, there is no other routine method used to reduce pain other than the administration of local anesthetic drops before the examination. Because of this situation, nurses apply various non-pharmacological methods to alleviate pain. These methods are; breast milk, sucrose use, oral dextrose use, non-nutritive sucking, positioning, listening to music and mother's voice. In the literature review; In a study evaluating the effectiveness of sucrose combination with non-nutritive sucking, they reported that pain was moderately reduced and more studies are needed. In another study (2015), it was concluded that topical anesthesia and oral dextrose were not effective in reducing pain in both groups. In a study comparing the effectiveness of breast milk and sucrose, it is recommended to use breast milk because of the rapid recovery of the baby after the ROP examination. In the comparison of the position, which is another non-pharmacological method, with the routine practice in the study conducted in 2019; It has been concluded that the frock position is more effective in relieving pain. In another study, it was stated that the mother's voice as music therapy also showed an analgesic effect and accelerated the recovery after the ROP examination. In the light of this information, when we look at the literature, no specific study was found in which a rain stick and The Happiest Baby music were used to reduce pain and increase the comfort level during the ROP examination. Therefore, this research will be carried out to determine the effect of different music played on the pain and comfort level of premature babies during the retinopathy examination.

ELIGIBILITY:
Inclusion Criteria:

* • Gestational age ≤34 weeks

  * Birth Weight ≤2000 grams
  * Preterm newborns with a corrected/postnatal age of 28-36 weeks at the time of examination
  * Having the baby's first ROP examination
  * Not giving sedative, opioid and anticonvulsant drugs before/during the examination
  * Parents do not have diagnosed mental or mental problems and agree to participate in the research.

Exclusion Criteria:

* Presence of a condition that prevents pain assessment (intracranial hemorrhage, neuromotor developmental retardation, etc.)

  * Oxygen requirement (nasal cannula, hood or incubator)
  * Having any congenital defect (eye, neurological) that may adversely affect the examination
  * Having a diagnosed hearing loss
  * Performing a different painful procedure at least one hour before the ROP
  * Being connected to a mechanical ventilator
  * Congenital hearing problems in family members

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Baby Information Form: | It will be applied when babies first arrive.
  This form consists of 6 questions including the baby's birth weight, birth week, current weight, corrected week, and delivery type.

SECONDARY OUTCOMES:
Premature Infant Pain Profile (PIPP) | Approximately 2 minutes of video will be recorded and measurement will be taken approximately in the first minute of the video and 2 minutes after the video.
  Pain assessment of preterm infants was performed with Premature Infant Pain Profile. The scale, which was developed by Stevens et al. in 1996 for 28-36 weeks preterms, is a multidimensional measurement tool with 7 sub-title evaluation criteria in the evaluation of acute pain in preterms (Gibbins et al., 2014). Turkish validity and reliability for all term and preterms were made by Derebent in 2007 within the scope of his master's thesis (Derebent, 2007). All sub-headings are scored between 0,1,2,3. According to the Turkish validity and reliability study of the scale, the highest score obtained from the scale is 21; 0-6 points indicate mild pain, 7-12 points indicate moderate pain, and 13-21 points indicate severe pain.

OTHER OUTCOMES:
Premature Baby Comfort Scale | Approximately 2 minutes of video will be recorded and measurement will be taken approximately in the first minute of the video and 2 minutes after the video.
  Ambuel et al. The comfort scale was developed by Monique et al. This scale was adapted to Turkish by Alemdar and Tüfekçi in 2015 by Alemdar and Tüfekçi. PBKO; It is a multidimensional scale used to evaluate behavioral and psychological comfort and pain. PBCS assesses 7 parameters such as Alertness, Calmness/Agitation, Respiratory Status (only with mechanical ventilation support) or Crying (not evaluated because it is scored only in children with spontaneous breathing), Physical Movement, Muscle Tone, Facial Movements, and Average Heart Rate. Accordingly, 35 indicates the lowest comfort score and 7 the highest. A high score on the scale indicates a low level of comfort. If the total score obtained is ≥17, it is the cut-off value of the scale, the limit value for the infant's comfort level, and indicates the need for an intervention to reduce pain.

CONTACTS AND LOCATIONS:
Overall Officials: Semra KÖSE, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilgeç, G. H., & Erol N. (2018). Epidemiology, Prevalence and Incidence in Retinopathy of Prematurity (Vol. 2, Issue 1). Chen, H. L., Chen, C. H., Wu, C. C., Huang, H. J., Wang, T. M., & Hsu, C. C. (2009). The Influence of Neonatal Intensive Care Unit Design on Sound Level. Pediatrics and Neonatology, 50(6), 270-274. https://doi.org/10.1016/S1875-9572(09)60076-0 Cohen, J. (2013). Statistical power analysis for the behavioral sciences. Routledge. Corrigan, M. J., Keeler, J. R., Miller, H. D., ben Khallouq, B. A., & Fowler, S. B. (2020). Music therapy and retinopathy of prematurity screening: using recorded maternal singing and heartbeat for post exam recovery. Journal of Perinatology, 40(12), 1780-1788. https://doi.org/10.1038/S41372-020-0719-9 Derebent, E. (2007). The Effect of Kangaroo Care on Reducing Pain During Invasive Procedures for Premature Babies. Dilli, D., Ilarslan, N. E. Ç., Kabataş, E. U., Zenciroǧlu, A., Şimşek, Y., & Okumuş, N. (2014). Oral sucrose and non-nutritive sucking goes some way to reducing pain during retinopathy of prematurity eye examinations. Acta Paediatrica (Oslo, Norway: 1992), 103(2). https://doi.org/10.1111/APA.12454 Dolgun, G. (2019). The Use of Pulse Oximetry in Defining Critical Congenital Heart Diseases and the Role of Midwife-Nurse. Journal of Education and Research in Nursing. https://doi.org/10.5222/head.2019.134 Gibbins, S., Stevens, B. J., Yamada, J., Dionne, K., Campbell-Yeo, M., Lee, G., Caddell, K., Johnston, C., & Taddio, A. (2014). Validation of the Premature Infant Pain Profile-Revised (PIPP-R). Early Human Development, 90(4), 189-193. https://doi.org/10.1016/J.EARLHUMDEV.2014.01.005 Koç, E., Yağmur, A., Prof, B., Özdek, S., & Ovali, F. (2021). Turkish Neonatology Society Turkish Ophthalmology Society Turkey Retinopathy of Prematurity Guideline 2021 Update. Küçük Alemdar, D., & Güdücü Tüfekci, F. (2015). The Reliability and Validity of the Premature Infant Comfort Scale's Turkish. Journal of Education and Research in Nursing. https://doi.org/10.5222/head.2015.142 Metres, O. (2014). Retinopathy of Prematurity from a Nursing Perspective. https://cms.galenos.com.tr/Uploads/Article_25271/European%20Archives%20of%20Medical%20Research-30-63-En.pdf Metreş, Ö., & Yıldız, S. (2019). Pain Management with ROP Position in Turkish Preterm Infants During Eye Examinations: A Randomized Controlled Trial. Journal of Pediatric Nursing, 49, e81-e89. https://doi.org/10.1016/J.PEDN.2019.08.013 Nesargi, S. v, Nithyanandam, S., Rao, S., Nimbalkar, S., & Bhat, S. (2015). Topical Anesthesia or Oral Dextrose for the Relief of Pain in Screening for Retinopathy of Prematurity: a Randomized Controlled Double-blinded Trial. https://doi.org/10.1093/tropej/fmu058 Parra, J., de Suremain, A., Berne Audeoud, F., Ego, A., & Debillon, T. (2017). Sound levels in a neonatal intensive care unit significantly exceeded recommendations, especially inside incubators. Acta Paediatrica, International Journal of Paediatrics, 106(12), 1909-1914. https://doi.org/10.1111/apa.13906 Sancak, S., Topçuoğlu, S., Çelik, G., Günay, M., & Karatekin, G. (2019). Frequency of Retinopathy of Prematurity and Evaluation of Risk Factors. Zeynep Kamil Medical Bulletin. https://doi.org/10.16948/zktipb.474762 Sun, X., Lemyre, B., Barrowman, N., & O'Connor, M. (2010). Pain management during eye examinations for retinopathy of prematurity in preterm infants: A systematic review. In Acta Paediatrica, International Journal of Paediatrics (Vol. 99, Issue 3, pp. 329-334). https://doi.org/10.1111/j.1651-2227.2009.01612.x Şener Taplak, A., & Erdem, E. (2017). A Comparison of Breast Milk and Sucrose in Reducing Neonatal Pain During Eye Exam for Retinopathy of Prematurity. Breastfeeding Medicine: The Official Journal of the Academy of Breastfeeding Medicine, 12(5), 305-310. https://doi.org/10.1089/BFM.2016.0122 Taplak, A. S., & Erdem, E. (2018). Pain Management in Examination for Retinopathy of Prematurity. In Journal of Health Sciences) (Vol. 27, Issue 2).